CLINICAL TRIAL: NCT02816710
Title: Different Conbercept Injection Methods in Treatment of Severe Proliferative Diabetic Retinopathy
Brief Title: Conbercept Injection in Treatment of Severe Proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Xi Shen, chief physician, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016062501
Record Dates: First submitted 2016-06-25; First posted 2016-06-28 (Estimated); Results first posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Proliferative Diabetic Retinopathy; Tractional Retinal Detachment
Keywords: Conbercept; Proliferative diabetic retinopathy; Silicone oil tamponade
MeSH Terms: interventions — KH902 fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IVC Preoperative group (Experimental): Conbercept injection before vitrectomy
  Interventions: Drug: Conbercept
- IVC Postoperative group (Experimental): Conbercept injection at the end of vitrectomy
  Interventions: Drug: Conbercept
- IVC Pre- and Post-operative group (Experimental): First conbercept injection before vitrectomy and second at the end of operation.
  Interventions: Drug: Conbercept

INTERVENTIONS:
Drug: Conbercept — Conbercept is a humanized soluble fusion protein which has a high binding affinity to the Fc region of human immunoglobulin G1 simultaneously. Prior clinical studies have demonstrated that intravitreal conbercept (IVC) inhibits the process of angiogenesis in vivo and in vitro, and has been recognized as a novel effective treatment strategy for neovascularization, providing an alternative treatment option for ophthalmologists.

SUMMARY:
To evaluate efficacy of different intravitreal Conbercept injection therapy in the treatment of severe proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
To assess the clinical effects of preoperative, intraoperative or preoperative combined with intraoperative intravitreal conbercept (IVC) injection in pars plana vitrectomy (PPV) with silicone oil tamponade for severe proliferative diabetic retinopathy (PDR). Methods. These patients were randomly assigned to three groups: Group 1 received an IVC injection 3 to 5 days before surgery; Group 2 received an IVC injection at the end of surgery; and Group 3 received an IVC injection 3 to 5 days before PPV as well as an IVC injection at the end of PPV. Follow-up examinations were performed for at least six months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of either sex aged ≥ 18 years.
2. Diagnosis of diabetes mellitus (type 1 or type 2);
3. Active proliferative diabetic retinopathy was clinically evident;
4. Study eyes required a vitrectomy and silicone oil tamponade due to vitreous hemorrhage with significant fibrous proliferation, tractional retinal detachment in the posterior pole or complicated retinal detachment, which can be detected by B-scan ultrasonography.
5. Ability to give informed consent.

Exclusion Criteria:

1. Coexistent ocular disease that may interfere with visual outcome;
2. Prior vitreoretinal surgery or anti-vascular endothelial growth factor (VEGF) pharmacotherapy in either eye;
3. A macula-involving retinal detachment for >6 months in the study eye;
4. Iris or angle neovascularization and neovascular glaucoma;
5. known allergy to any components of conbercept formulation
6. severe external ocular infection;
7. pregnancy or current oral contraceptive intake;
8. usage of anticoagulant or antiplatelet therapy;
9. preoperative or postoperative poor diabetes control [serum hemoglobin A1c (HbA1c) >11.0%];
10. uncontrolled systemic diseases, such as hypertension, cardiac diseases or presenting abnormal coagulation-associated blood diseases;
11. <6 months of follow-up post initial surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xi Shen, PhD, Study Director — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed in the department of Ophthalmology, Ruijin Hospital, affiliated with Shanghai Jiaotong University School of Medicine, between July 2016 and September 2017.
Groups:
- IVC Preoperative Group: Patients in this group received an intravitreal conbercept (IVC) injection 3 to 5 days before surgery.
- IVC Postoperative Group: Patients in this group received an IVC injection at the end of surgery.
- IVC Pre- and Post-operative Group: Patients in this group received an IVC injection 3 to 5 days before PPV as well as an IVC injection at the end of pars plana vitrectomy (PPV).
Period: Overall Study
Arm/Group | IVC Preoperative Group | IVC Postoperative Group | IVC Pre- and Post-operative Group
Started | 38 | 38 | 36
Completed | 34 | 35 | 29
Not Completed | 4 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVC Preoperative Group | IVC Postoperative Group | IVC Pre- and Post-operative Group | Total
Number analyzed (Participants) | 34 | 35 | 29 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.76 (13.47) | 53.97 (14.76) | 52.55 (14.62) | 52.44 (14.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 13 | 52
  Male | 14 | 16 | 16 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Hypertension [Count of Participants; unit: Participants] | 15 | 17 | 13 | 45
HbA1c at time of surgery [Mean (Standard Deviation); unit: %] | 7.12 (1.52) | 7.59 (1.36) | 7.88 (1.26) | 7.51 (1.41)
Type 1 diabetes [Count of Participants; unit: Participants] | 3 | 2 | 3 | 8
Duration of diabetes (years) [Mean (Standard Deviation); unit: years] | 14.50 (5.16) | 12.86 (5.23) | 12.66 (5.24) | 13.37 (5.22)
Study eye (right eye) [Number; unit: eyes] | 21 | 17 | 16 | 54
Previous history of pan-retinal photocoagulation (PRP) [Count of Participants; unit: Participants] | 11 | 15 | 13 | 39
LogMAR Best Corrected Visual Acuity (BCVA) [Mean (Standard Deviation); unit: LogMAR] | 1.95 (0.43) | 1.97 (0.37) | 1.98 (0.44) | 1.96 (0.41)
Lens status (pseudophakic) [Count of Participants; unit: Participants] | 4 | 3 | 7 | 14
Preoperative iris neovascularization [Count of Participants; unit: Participants] | 2 | 3 | 2 | 7
Extent of vitreoretinal adhesion grade [Count of Participants; unit: Participants] — The extent of vitreoretinal adhesion was assessed based on a previous grading system: Grade 0, without any adhesion; Grade 1, focal adhesion in less than 3 sites; Grade 2, broad adhesion in more than 1 site or adhesion at the disc, macular, or vascular arcade; Grade 3, vitreoretinal adhesion extending to the periphery. Grade 3 is considered to be the worst outcome.
  Participants
    3 | 9 | 10 | 17 | 36
    2 | 11 | 10 | 8 | 29
    1 | 14 | 15 | 4 | 33
    0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Best-corrected Visual Acuity
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- IVC Pre- and Post-operative Group: Patients in this group received an IVC injection 3 to 5 days before PPV as well as an IVC injection at the end of PPV.
Arm/Group | IVC Preoperative Group | IVC Postoperative Group | IVC Pre- and Post-operative Group
Number analyzed (Participants) | 34 | 35 | 29
LogMAR | 1.25 (0.45) | 1.29 (0.46) | 1.16 (0.44)

2. Primary Outcome: Duration of Surgery
Description: To evaluate the influence of these three methods to the final duration of surgery. We carefully estimated the time of the vitrectomy from insertion to extraction of the 23-gauge three-port trocars.
Time Frame: during the operation time
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | IVC Preoperative Group | IVC Postoperative Group | IVC Pre- and Post-operative Group
Number analyzed (Participants) | 34 | 35 | 29
minutes | 55.41 (11.24) | 67.66 (15.15) | 57.86 (13.23)

3. Primary Outcome: Intraoperative Bleeding
Description: The grading criteria for intraoperative bleeding: Grade 1, spontaneous cessation of minor bleeding or bleeding that stopped by transient elevation of perfusion pressure; Grade 2, moderate bleeding requiring endodiathermy or broad blood clots formed far away from the bleeding site; Grade 3, thick blood clots exceeding half of the posterior pole or affecting the operation field.
Time Frame: Time between the insertion and extraction of three 23-gauge vitrectomy ports
Measure: Count of Participants; unit: Participants
Arm/Group | IVC Preoperative Group | IVC Postoperative Group | IVC Pre- and Post-operative Group
Number analyzed (Participants) | 34 | 35 | 29
Participants
  Grade 1 | 15 | 7 | 12
  Grade 2 | 12 | 16 | 11
  Grade 3 | 7 | 12 | 6

4. Secondary Outcome: Postoperative Preretinal Blood
Description: The grading criteria for postoperative preretinal blood: Grade 1, isolated blood clots within 10 disk area but without covering the posterior pole; Grade 2, broad blood clots exceeding 10 disk area regardless of involvement of the posterior pole; Grade 3, broad blood clots exceeding 10 disk area as well as involving the posterior pole. Maximal extent of preretinal blood within 1 week postoperatively was used for grading the extent of hemorrhage.
Time Frame: postoperatively, up to 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | IVC Preoperative Group | IVC Postoperative Group | IVC Pre- and Post-operative Group
Number analyzed (Participants) | 34 | 35 | 29
Participants
  Grade 1 | 14 | 15 | 17
  Grade 2 | 11 | 11 | 8
  Grade 3 | 9 | 9 | 4

5. Secondary Outcome: Reabsorption Time of Blood
Description: To monitor the reabsorption time of preretinal blood.
Time Frame: follow up period, up to an average of 6 months after the operation
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IVC Preoperative Group | IVC Postoperative Group | IVC Pre- and Post-operative Group
Number analyzed (Participants) | 34 | 35 | 29
days | 11.24 (4.33) | 12.23 (6.19) | 10.10 (4.07)

6. Secondary Outcome: Recurrent Vitreous Hemorrhage
Description: Recurrent vitreous hemorrhage(VH) was referred to any new episode of VH occurring after one week postoperatively, dividing into early stage (≤ 4 weeks) and late stage (> 4 weeks).
Time Frame: follow up period, up to an average of 6 months after the operation
Measure: Count of Participants; unit: Participants
Arm/Group | IVC Preoperative Group | IVC Postoperative Group | IVC Pre- and Post-operative Group
Number analyzed (Participants) | 34 | 35 | 29
Participants
  early vitreous hemorrhage | 6 | 7 | 2
  late vitreous hemorrhage | 5 | 3 | 2
  no vitreous hemorrhge | 23 | 25 | 25

7. Secondary Outcome: Frequency of Intraoperative Electrocoagulation
Description: The number of times electrocoagulation, which was used to stop bleeding, was carefully counted.
Time Frame: during the operation time
Measure: Mean (Standard Deviation); unit: events
Groups:
- Group 1: Group 1 received an intravitreal conbercept (IVC) injection 3 to 5 days before surgery.
- Group 2: Group 2 received an IVC injection at the end of surgery.
- Group 3: Group 3 received an IVC injection 3 to 5 days before PPV as well as an IVC injection at the end of PPV.
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 34 | 35 | 29
events | 1.73 (1.26) | 3.00 (1.14) | 1.34 (0.81)

8. Secondary Outcome: Number of Participants With Neovascular Glaucoma (NVG)
Time Frame: follow up period, up to an average of 6 months after the operation
Measure: Count of Participants; unit: Participants
Arm/Group | IVC Preoperative Group | IVC Postoperative Group | IVC Pre- and Post-operative Group
Number analyzed (Participants) | 34 | 35 | 29
Participants | 4 | 5 | 2

9. Secondary Outcome: Recurrent Retinal Detachment
Time Frame: follow up period, up to an average of 6 months after the operation
Measure: Count of Participants; unit: Participants
Arm/Group | IVC Preoperative Group | IVC Postoperative Group | IVC Pre- and Post-operative Group
Number analyzed (Participants) | 34 | 35 | 29
Participants | 4 | 5 | 3

10. Secondary Outcome: Need for Reoperation
Description: due to recurrent retinal detachment or unclear vitreous hemorrhage
Time Frame: follow up period, up to an average of 6 months after the operation
Measure: Count of Participants; unit: Participants
Arm/Group | IVC Preoperative Group | IVC Postoperative Group | IVC Pre- and Post-operative Group
Number analyzed (Participants) | 34 | 35 | 29
Participants | 11 | 9 | 6

ADVERSE EVENTS:
Time Frame: 6 months
Description: Systemic adverse events such as heart failure, myocardial infarction or acute cerebrovascular diseases and ocular adverse events like endophthalmitis or ocular toxicity were observed in all participants.
Arm/Group | IVC Preoperative Group | IVC Postoperative Group | IVC Pre- and Post-operative Group
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35 | 0/29
Other Adverse Events (participants affected / at risk) | 0/34 | 0/35 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT02816710/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT02816710/SAP_001.pdf